CLINICAL TRIAL: NCT01201161
Title: The Effect of Intravitreous Ranibizumab on Intra-Operative Bleeding During Pars Plana Vitrectomy for Diabetic Traction Retinal Detachment
Brief Title: Ranibizumab for Diabetic Traction Retinal Detachment
Acronym: RANITRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RANITRA
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-01

CONDITIONS: Diabetic Retinopathy; Retinal Detachment
Keywords: Diabetic Retinopathy; Retinal detachment; Vitreous Hemorrhage; Preoperative Ranibizumab; pars plana vitrectomy
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Detachment; Vitreous Hemorrhage | interventions — Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RANI/PPV (Experimental): Preoperative intravitreal ranibizumab and pars plana vitrectomy
  Interventions: Drug: Ranibizumab
- PPV (Placebo Comparator): Sham injection and pars plana vitrectomy
  Interventions: Other: Sham injection

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal injection of ranibizumab 0.05 ml (0.5 mg) one week before pars plana vitrectomy
  Other Names: Lucentis
  Arms: RANI/PPV
Other: Sham injection — Simulation of intravitreal injection one week before pars plana vitrectomy
  Arms: PPV

SUMMARY:
The purpose of this study was to assess the effect of ranibizumab in reducing intraoperative vitreous haemorrhage during pars plana vitrectomy, thus facilitating surgery and improving its anatomical and functional results in patients with advanced proliferative diabetic retinopathy and traction retinal detachment.

ELIGIBILITY:
Inclusion Criteria:

* Macular traction retinal detachment lasting three months or less secondary to diabetic retinopathy.

Exclusion Criteria:

* Massive vitreous hemorrhage preventing from detailed posterior pole examination;
* Previous intra-ocular surgery other than cataract surgery
* Hemodialysis, known bleeding disorders or use of anticoagulants drugs other than aspirin
* Prothrombin time, partial thromboplastin time or platelet count without normal limits
* History of previous thromboembolic events

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
amount of intraoperative intra-ocular bleeding | one week
  amount of intra-ocular bleeding that occurred during pars plana vitrectomy

SECONDARY OUTCOMES:
visual acuity | 12 weeks
  ETDRS best corrected visual acuity at 12 weeks after pars plana vitrectomy

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Jorge, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo, Ribeirão Preto, São Paulo, Brazil